CLINICAL TRIAL: NCT00955942
Title: A Phase I Blinded, Randomized Feasibility Trial of Dietary Flaxseed Administration in Non-Small Cell Lung Cancer Patients Receiving Definitive Thoracic Chemoradiotherapy
Brief Title: Flaxseed Supplement in Treating Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Undergoing Chemotherapy and Radiation Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000644401; UPCC-07507; IRB# 806733
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer; Radiation Toxicity
Keywords: radiation toxicity; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Radiation Injuries; Carcinoma, Non-Small-Cell Lung | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients consume flaxseed muffins once or twice daily beginning on the first day of radiotherapy and continuing for up to 9-10 weeks.
  Interventions: Dietary Supplement: flaxseed
- Arm II (Placebo Comparator): Patients consume placebo muffins once or twice daily beginning on the first day of radiotherapy and continuing for up to 9-10 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: flaxseed — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Flaxseed may help protect normal cells from the side effects of radiation therapy.

PURPOSE: This randomized phase I trial is studying the side effects of flaxseed supplement in treating patients with locally advanced or metastatic non-small cell lung cancer undergoing chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility of dietary flaxseed (FS) supplementation in patients undergoing definitive chemoradiotherapy for locally advanced or metastatic non-small cell lung cancer.
* To collect toxicity and tolerability data on dietary FS supplementation during definitive chemoradiotherapy.

Secondary

* To validate urinary and serum markers of oxidative stress and FS lignan levels as surrogates of the bioavailability of FS in these patients.
* To determine if a dose response to daily ingestion of 20 g or 40 g of FS can be observed in plasma lignan levels and urinary markers of oxidative stress.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients consume flaxseed muffins once or twice daily beginning on the first day of radiotherapy and continuing for up to 9-10 weeks.
* Arm II: Patients consume placebo muffins once or twice daily beginning on the first day of radiotherapy and continuing for up to 9-10 weeks.

Blood and urine samples are collected periodically for biomarker studies.

After completion of study treatment, patients are followed up for 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer

  * Locally advanced or metastatic disease
* Requires definitive thoracic and mediastinal radiotherapy with concurrent chemotherapy

  * Total planned radiation dose to gross disease 60-80 Gy

PATIENT CHARACTERISTICS:

* No diagnosis of disease of the gastrointestinal (GI) system, liver, or kidneys that could result in altered metabolism or excretion of the study medication (e.g., history of major GI tract surgery, gastrectomy, gastrostomy, or bowel resection)
* No history of chronic GI disorders (e.g., ulcerative colitis, regional enteritis, or GI bleeding)
* No known hypersensitivity to flaxseed or any of its metabolites or to wheat products

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* See Patient Characteristics
* More than 14 days since prior and no concurrent investigational drugs
* More than 14 days since prior and no concurrent amifostine or Mucomyst (N-acetylcysteine)
* No prior thoracic radiotherapy
* No prior or other concurrent flaxseed, flax-containing products, soybeans, or soy-containing products
* No other concurrent dietary supplements, such as herbals or botanicals

  * Vitamins or multivitamins, including calcium and vitamin D, are allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12; Primary Completion 2012-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of dietary flaxseed (FS) supplementation
Toxicity and tolerability of dietary FS supplementation during chemoradiotherapy

SECONDARY OUTCOMES:
Measures of biomarkers of oxidative stress
Measures of serum levels of FS metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States